CLINICAL TRIAL: NCT03468543
Title: A Study Designed to Determine the Gastro-Retentive and Modified Release Properties of Memantine Hydrochloride (HCl) Prototype Capsule Formulations in Healthy Subjects
Brief Title: Study Determining Gastric-Retentive and Modified Release Properties of Prototype Capsules in Healthy Subjects
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Per protocol stopping rules
Sponsor: Lyndra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: QCL117924; 2017-000982-61 (EudraCT Number)
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-08

CONDITIONS: Gastric Retention; Healthy
MeSH Terms: interventions — Memantine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Subjects will receive an oral administration of 50 mg of Memantine HCl prototype capsule formulation A; then formulation B; following each administration MRI will be performed for up to 14 days
  Interventions: Drug: Memantine Hydrochloride MR Prototype Capsule Formulation A; Drug: Memantine Hydrochloride MR Prototype Capsule Formulation B; Procedure: Magnetic Resonance Imaging
- Cohort 2 (Experimental): Subjects will receive an oral administration of 50 mg of Memantine HCl prototype capsule formulation C; then formulation D; following each administration MRI will be performed for up to 14 days
  Interventions: Drug: Memantine Hydrochloride MR Prototype Capsule Formulation C; Drug: Memantine Hydrochloride MR Prototype Capsule Formulation D; Procedure: Magnetic Resonance Imaging
- Cohort 3 (Experimental): Subjects will receive an oral administration of 50 mg of Memantine HCl prototype capsule formulation E; followed by MRI for up to 14 days
  Interventions: Drug: Memantine Hydrochloride MR Prototype Capsule Formulation E; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Memantine Hydrochloride MR Prototype Capsule Formulation A — Memantine HCl MR capsule formulation will be administered orally in a single dose
  Other Names: Memantine HCl Capsule Formulation A (50 mg)
  Arms: Cohort 1
Drug: Memantine Hydrochloride MR Prototype Capsule Formulation B — Memantine HCl MR capsule formulation will be administered orally in a single dose
  Other Names: Memantine HCl Capsule Formulation B (50 mg)
  Arms: Cohort 1
Drug: Memantine Hydrochloride MR Prototype Capsule Formulation C — Memantine HCl MR capsule formulation will be administered orally in a single dose
  Other Names: Memantine HCl Capsule Formulation C (50 mg)
  Arms: Cohort 2
Drug: Memantine Hydrochloride MR Prototype Capsule Formulation D — Memantine HCl MR capsule formulation will be administered orally in a single dose
  Other Names: Memantine HCl Capsule Formulation D (50 mg)
  Arms: Cohort 2
Drug: Memantine Hydrochloride MR Prototype Capsule Formulation E — Memantine HCl MR capsule formulation will be administered orally in a single dose
  Other Names: Memantine HCl Capsule Formulation E (50 mg)
  Arms: Cohort 3
Procedure: Magnetic Resonance Imaging — MRI will be performed on specified days according to protocol
  Other Names: MRI

SUMMARY:
To assess how long modified release (MR) memantine hydrochloride prototype capsule formulations stay in the stomach as determined by magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
This is a single center, open-label, single dose, 5-period study in 24 healthy male and female subjects, with an optional Period 6, if required. It is expected the study will be executed in 3 cohorts of 8 subjects, with each cohort participating in up to 2 study periods (total of up to 6 study periods). Cohort 3 may be conducted in parallel with Cohort 2.

Subjects will be dosed in a sequential manner, as appropriate. Each subject will be administered up to 2 regimens (2 different prototype capsule formulations) across 2 study periods. There will be a minimum 35-day interval between each dose administration.

Subjects will have an MRI scan performed on Days 2, 4, 7, 10 and 14 of each period to assess the gastric retentive properties of the formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects.
2. Body mass index of 18.0 to 32.0 kg/m2.
3. Subjects must demonstrate their ability to swallow a test capsule at screening.
4. Must provide written informed consent.

Exclusion Criteria:

1. Subjects who have received any investigational medicinal product in a clinical research study within the previous 3 months.
2. Subjects who have previously been enrolled in this study.
3. History of any drug or alcohol abuse in the past 2 years.
4. Current smokers and those who have smoked within the last 12 months.
5. Individuals with clinically significant medical history relating to the gastrointestinal tract and potential for complications, thereof
6. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
7. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
8. Individuals with contraindication to MRI imaging.

Other protocol defined criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MBChB, DRCOG, Study Director — Quotient Clinical
Locations (1):
- Quotient Sciences (formerly Quotient Clinical), Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Subjects will receive an oral administration of 50 mg of Memantine HCl prototype capsule formulation A; then formulation B; following each administration MRI will be performed for up to 14 days
  Memantine Hydrochloride MR Prototype Capsule Formulation A: Memantine HCl MR capsule formulation will be administered orally in a single dose
  Memantine Hydrochloride MR Prototype Capsule Formulation B: Memantine HCl MR capsule formulation did NOT get administered
  Magnetic Resonance Imaging: MRI will be performed on specified days according to protocol
Period: Overall Study
Arm/Group | Cohort 1
Started | 3
Completed | 0
Not Completed | 3
Not completed — Protocol stopping rules met | 3

BASELINE CHARACTERISTICS:
Population: Cohorts 2 and 3 were not executed, as the study was stopped during Cohort 1
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (12.3) |  |  | 33.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  |  | 0
  Male | 3 |  |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 1 |  |  | 1
  White | 2 |  |  | 2
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Gastric Retention by Magnetic Resonance Imaging (MRI)
Description: Number of Participants with Gastric Retention by Magnetic Resonance Imaging (MRI), as measured after dosing
Time Frame: 7 Days
Population: Subjects who completed dosing and at least one MRI assessment after dosing
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected for five weeks after each dose of study drug.
Description: Additional information:
  Adverse events were collected for five weeks after each dose of study drug in Cohort 1 only. Cohorts 2 and 3 were not performed as the study was stopped, therefore the number of participants at risk for AE's (all types) is zero.
Groups:
- Cohort 1: Subjects will receive an oral administration of 50 mg of Memantine HCl prototype capsule formulation A; then formulation B; following each administration MRI will be performed for up to 14 days
  Memantine Hydrochloride MR Prototype Capsule Formulation A: Memantine HCl MR capsule formulation will be administered orally in a single dose
  Memantine Hydrochloride MR Prototype Capsule Formulation B: Memantine HCl MR capsule formulation was NOT administered
  Magnetic Resonance Imaging: MRI will be performed on specified days according to protocol
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3)
foreign body (Injury, poisoning and procedural complications) | 1 (1) — medication stuck in throat
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3)
presyncope (Nervous system disorders) | 1 (1)
crying (General disorders) | 1 (1)
non-cardiac chest pain (General disorders) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1)
abdominal discomfort (Gastrointestinal disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (4)
dysphagia (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was prematurely ended after the dosing of three subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT03468543/Prot_SAP_000.pdf